CLINICAL TRIAL: NCT02344810
Title: A Phase I and Randomized Phase II Double Blinded Placebo Controlled Study of mFOLFOX6 +/- AMG 337 in the First Line Treatment of Patients With Her2/Neu Negative and High MET Expressing Advanced Gastric and Esophageal Adenocarcinoma
Brief Title: C-Met Inhibitor AMG 337, Oxaliplatin, Leucovorin Calcium, and Fluorouracil in Treating Patients With Advanced Stomach or Esophageal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study did not open to accrual. No start date and no completion dates.
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); ECOG-ACRIN Cancer Research Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA2132; NCI-2014-01315 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2132 (Other: ECOG-ACRIN Cancer Research Group); EA2132 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Gastroesophageal Junction; Diffuse Adenocarcinoma of the Stomach; Gastrointestinal Cancer; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Stage IIIA Esophageal Cancer; Stage IIIA Gastric Cancer; Stage IIIB Esophageal Cancer; Stage IIIB Gastric Cancer; Stage IIIC Esophageal Cancer; Stage IIIC Gastric Cancer; Stage IV Esophageal Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Gastrointestinal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms | interventions — AMG 337; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (AMG 337, mFOLFOX6) (Experimental): Patients receive c-Met inhibitor AMG 337 PO QD on days 1-28; and oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46-48 hours on days 1 and 15.
  Interventions: Drug: c-Met inhibitor AMG 337; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm B (placebo, mFOLFOX6) (Active Comparator): Patients receive placebo PO QD on days 1-28; and oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46-48 hours on days 1 and 15.
  Interventions: Other: placebo; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: c-Met inhibitor AMG 337 — Given PO
  Other Names: AMG 337; AMG337
  Arms: Arm A (AMG 337, mFOLFOX6)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm B (placebo, mFOLFOX6)
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This partially randomized phase I/II trial studies the side effects and best dose of c-Met inhibitor AMG 337 when given together with oxaliplatin, leucovorin calcium, and fluorouracil and to see how well they work in treating patients with stomach or esophageal cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment. C-Met inhibitor AMG 337 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as, oxaliplatin, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving c-Met inhibitor AMG 337 with oxaliplatin, leucovorin calcium, and fluorouracil may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity of combination therapy with AMG 337 (c-Met inhibitor AMG 337) and mFOLFOX6 (oxaliplatin, leucovorin calcium, and fluorouracil) chemotherapy in patients with advanced or metastatic gastrointestinal (GI) cancers. (Phase I) II. To determine the dose of AMG 337 to be used in combination with mFOLFOX6 chemotherapy in the phase II portion of the trial. (Phase I) III. To determine the pharmacokinetics of AMG 337 in combination with mFOLFOX6. (Phase I) IV. To determine if the addition of AMG 337 to mFOLFOX6 chemotherapy improves median progression-free survival (PFS) in the first line treatment of patients with human epidermal growth factor receptor 2 (Her2Neu) negative and high c-met proto-oncogene (MET) expressing advanced esophagogastric and gastroesophageal junction (GEJ) adenocarcinoma. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the addition of AMG 337 to mFOLFOX6 chemotherapy and also to evaluate the placebo/mFOLFOX6 chemotherapy combination in the first line treatment of patients with Her2Neu negative and high c-MET expressing advanced esophagogastric and GEJ adenocarcinoma, with regards to overall survival (OS). (Phase II) II. To evaluate the addition of AMG 337 to mFOLFOX6 chemotherapy and also to evaluate the placebo/mFOLFOX6 chemotherapy combination in the first line treatment of patients with Her2Neu negative and high c-MET expressing advanced esophagogastric and GEJ adenocarcinoma, with regards to response rate and disease control rate. (Phase II) III. To evaluate the addition of AMG 337 to mFOLFOX6 chemotherapy and also to evaluate the placebo/mFOLFOX6 chemotherapy combination in the first line treatment of patients with Her2Neu negative and high c-MET expressing advanced esophagogastric and GEJ adenocarcinoma, with regards to toxicity rates. (Phase II) IV. To evaluate the addition of AMG 337 to mFOLFOX6 chemotherapy and also to evaluate the placebo/mFOLFOX6 chemotherapy combination in the first line treatment of patients with Her2Neu negative and high c-MET expressing advanced esophagogastric and GEJ adenocarcinoma, with regards to time to development of new metastasis. (Phase II) V. To evaluate the addition of AMG 337 to mFOLFOX6 chemotherapy and also to evaluate the placebo/mFOLFOX6 chemotherapy combination in the first line treatment of patients with Her2Neu negative and high c-MET expressing advanced esophagogastric and GEJ adenocarcinoma, with regards to evaluation of MET amplification. (Phase II) VI. To evaluate the addition of AMG 337 to mFOLFOX6 chemotherapy and also to evaluate the placebo/mFOLFOX6 chemotherapy combination in the first line treatment of patients with Her2Neu negative and high c-MET expressing advanced esophagogastric and GEJ adenocarcinoma, with regards to evaluation of MET amplification and MET expression as determined by DAKO immunohistochemistry (IHC) for comparison to Ventana IHC. (Phase II) VII. To evaluate the addition of AMG 337 to mFOLFOX6 chemotherapy and also to evaluate the placebo/mFOLFOX6 chemotherapy combination in the first line treatment of patients with Her2Neu negative and high c-MET expressing advanced esophagogastric and GEJ adenocarcinoma, with regards to a retrospective re-evaluation of the cutpoint used by the computer algorithm for c-MET IHC to assess its ability to distinguish responding versus non-responding patients will be undertaken in this population, so that a potentially more optimal cutpoint to define high c-MET tumors in patients can be identified. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of c-Met inhibitor AMG 337 followed by a phase II study.

PHASE I: Patients receive c-Met inhibitor AMG 337 orally (PO) once daily (QD) on days 1-28; and oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46-48 hours on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive c-Met inhibitor AMG 337 PO QD on days 1-28; and oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46-48 hours on days 1 and 15.

ARM B: Patients receive placebo PO QD on days 1-28; and oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46-48 hours on days 1 and 15.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study within 48 hours prior to randomization to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study therapy and for 3 months after the last dose of AMG 337 plus mFOLFOX6 chemotherapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; should a man impregnate or suspect that he has impregnated a woman while participating in this study, he should inform his treating physician immediately
* Patients must NOT have a known immediate or delayed hypersensitivity reaction to drugs chemically related to fluorouracil, platins or their excipients nor have a known history of dihydropyrimidine dehydrogenase (DPD) deficiency
* Patients must be able to swallow tablets whole
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional upper limit of normal (ULN) or =< 5 X ULN if the patient has liver metastases
* Creatinine =< 1.5 X institutional ULN or creatinine clearance >= 50 mL/min for patients with creatinine levels above institutional normal
* Patients must NOT be taking current medications or substances that are inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)
* Patients with known human immunodeficiency virus (HIV) are not eligible if cluster of differentiation (CD)4 count is =< 200 cell/mm^3 or if receiving antiretroviral therapy
* Patients must not have a pre-existing > grade 1 (Common Terminology Criteria for Adverse Events version 4 [CTCAEv4]) motor or sensory neuropathy
* Patients must not have an uncontrolled infection, active hepatic, biliary disease or other uncontrolled intercurrent illnesses including, but not limited to: uncontrolled ascites, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/addictive disorders that would limit compliance with study requirements
* PHASE I:
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria within 4 weeks prior to registration; patients must not have clinical or radiographic evidence of brain metastasis
* Patients must have histologically or cytologically confirmed adenocarcinoma originating from anywhere in the gastrointestinal tract
* Patients must have progression on standard therapies, for which effective therapy is not available (or patients are not a candidate for or are intolerant of such therapies)
* Patients must NOT have previous or concurrent malignancy; exceptions are made for patients who meet any of the following conditions:

  * Non-melanoma skin cancer, in situ cervical cancer, breast cancer in situ, or superficial bladder cancer (noninvasive papillary carcinoma or carcinoma in situ)
  * Prior malignancy completely excised or removed and patient has been continuously disease free for > 5 years from registration
* Patients may have received prior surgery or radiotherapy if > 4 weeks prior to registration and patient does not have any unresolved or unstable serious toxicity
* Patients must not be receiving an investigational agent concurrently and must not have received any other investigational agents within 4 weeks prior to randomization
* PHASE II:
* Patients must have measurable disease by RECIST 1.1 criteria within 4 weeks prior to registration to Step 0; patients must not have clinical or radiographic evidence of brain metastasis because of their poor prognosis
* Patient disease status must be as follows:

  * Adenocarcinoma or poorly differentiated carcinoma of the stomach, esophagus or gastroesophageal (GE) junction
  * Histologically or cytologically confirmed Her2/neu negative cancer prior to pre-registration; Her2/neu status must be determined by a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory
  * Locally advanced or metastatic disease that is inoperable and not amenable to curative therapy; linitis plastica is permitted
  * Patient must NOT have gastric carcinoid, sarcomas or squamous cell carcinoma
* Patients may have received prior surgery or radiotherapy if > 4 weeks prior to registration to Step 0 and patient does not have any unresolved or unstable serious toxicity
* Patients must NOT have previous or concurrent malignancy; exceptions are made for patients who meet any of the following conditions:

  * Non-melanoma skin cancer, in situ cervical cancer, breast cancer in situ, or superficial bladder cancer (noninvasive papillary carcinoma or carcinoma in situ)
  * Prior malignancy completely excised or removed and patient has been continuously disease free for > 5 years from registration to Step 0
* Patients must not be receiving an investigational agent concurrently and must not have received any other investigational agents within 4 weeks prior to registration to Step 0
* Patient may not have received prior chemotherapy for advanced disease or prior oxaliplatin or anti-MET therapy
* Previous neo-adjuvant or adjuvant treatment is allowed provided that it was discontinued >= 6 months prior to registration to Step 0
* Patients must have paraffin-embedded tumor specimen available for submission for central determination of MET expression status

  * NOTE: it is recommended that patients not be pre-registered until the required tumor specimens are on hand and ready for submission; if submission of tissue will be submitted more than 5 working days after pre-registration, immediately notify the receiving laboratory
* Patients must have had MET expression status determined by the Immunohistochemistry Laboratory and Image Analysis Laboratory in the Department of Pathology of The University of Texas MD Anderson Cancer Center in Houston: the report from the central laboratory indicates tumor tissue has MET

  * NOTE: for this protocol, 'MET High' will be defined as: >= 50% tumor cells with a staining intensity of 2+ or 3+ in IHC utilizing the CONFIRM anti-total MET, SP44, rabbit monoclonal primary antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-06; Primary Completion 2015-03-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of c-Met inhibitor AMG 337, defined as the highest dose level at which < 33% of 6 patients experience a dose limiting toxicity graded according to CTCAE v.4 (Phase I) | 28 days
Progression-free survival (Phase II) | Up to 2 years
  The study will have 90% power to detect the above improvement in PFS using a one-sided 0.10 level log rank test.

SECONDARY OUTCOMES:
Overall survival (Phase II) | Up to 2 years
Response rate (Phase II) | Up to 2 years
Disease control rate (Phase II) | Up to 2 years
Incidence of toxicity graded according to CTCAE v.4 (Phase II) | Up to 2 years
  The study will have at least 83% power to detect an absolute differences of 26% or more (e.g. 64% versus 38% true toxicity rates) between the two arms for any given adverse event, using a one-sided 5% level Fisher's exact test.
Time to development of new metastasis (Phase II) | Up to 2 years
Evaluation of MET amplification via fluorescence in situ hybridization (FISH) (Phase II) | Up to 2 years
Evaluation of MET amplification and MET expression as determined by DAKO IHC (Phase II) | Up to 2 years
  Comparison of DAKO IHC to Ventana IHC and comparison of amplification by FISH to overexpression by Ventana IHC amongst all pre-registered patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Rajdev, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States